CLINICAL TRIAL: NCT02528331
Title: Cognitive Behavioral Strategies and Transcranial Magnetic Stimulation in Obsessive-Compulsive Disorder: Open Label Study
Acronym: CBT-TMS
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: PI has left Duke
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: Pro00047168
Record Dates: First submitted 2015-08-17; First posted 2015-08-19 (Estimated); Results first posted 2017-02-09 (Estimated); Last update posted 2017-02-09 (Estimated); Status verified 2016-11

CONDITIONS: Obsessive Compulsive Disorder (OCD)
Keywords: Transcranial magnetic stimulation (TMS); Cognitive behavioral therapy (CBT)
MeSH Terms: conditions — Obsessive-Compulsive Disorder | interventions — Transcranial Magnetic Stimulation; Cognitive Behavioral Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- rTMS and Cognitive Behavior Therapy (Experimental)
  Interventions: Device: Transcranial magnetic stimulation; Behavioral: Cognitive behavioral therapy

INTERVENTIONS:
Device: Transcranial magnetic stimulation
Behavioral: Cognitive behavioral therapy

SUMMARY:
The purpose of this study is to evaluate the effectiveness of repetitive TMS (rTMS) delivered simultaneously with elements of cognitive behavioral therapy/exposure-response prevention (CBT/ERP) in adult subjects (greater or equal to 18 years old) with obsessive-compulsive disorder (OCD). This is an open label study that involves standard of care for OCD (CBT) and an investigational treatment modality (TMS). The investigators will compare the Yale-Brown Obsessive Compulsive Scale (YBOCS) scores before and after treatment to quantify clinical improvement. The side effects from TMS include, but are not limited to, headache, seizure, and general pain. CBT has minimal side effects other than mental discomfort during the exposure sessions. For safety concerns, pregnant women and subjects with seizure-related history will be excluded as well as other indicated conditions in the details protocol.

ELIGIBILITY:
Inclusion Criteria

Subjects must meet all of the following inclusion criteria to qualify for enrollment into the study:

1. All subjects will be 18 - 65 years of age.
2. Obsessive-compulsive disorder:

   * Subjects will meet the DSM-IV primary diagnosis of obsessive-compulsive
   * Y-BOCS total score > 16
3. Subjects are willing and able to adhere to the intensive treatment schedule and all required study visits.

Exclusion Criteria

Subjects will be excluded from study participation if one of the following exclusion criteria applies:

1. Subjects are unable or unwilling to give informed consent.
2. No exclusion criteria for comorbid DSM diagnosis.
3. Subjects with a clinically defined neurological disorder that caused significant safety concern to receive TMS treatment, including, but not limited to:

   * Any condition likely to be associated with increased intracranial pressure.
   * Space occupying brain lesion.
   * Any history of seizure EXCEPT those therapeutically induced by ECT (childhood febrile seizures are acceptable and these subjects may be included in the study).
   * History of stroke.
   * Transient ischemic attack within two years.
   * Cerebral aneurysm.
   * Dementia.
   * Mini Mental Status Exam (MMSE-2) score of <24.
   * Parkinson's disease.
   * Huntington's disease.
   * Multiple sclerosis.
   * Increased risk of seizure for any reason, including prior diagnosis of increased intracranial pressure (such as after large infarctions or trauma), or currently taking medication that lowers the seizure threshold. Medications that lower the seizure threshold are included in the Prohibited Concomitant Medication (Section 5.8).
4. Subjects with any of the following treatment histories:

   * TMS treatment within 6 months prior to the screening visit.
   * Lifetime history of treatment with Deep Brain Stimulation
   * Use of any investigational drug or device within 4 weeks of the randomization visit.
   * If participating in psychotherapy, must have been in stable treatment for at least 2 months prior to entry into the study, with no anticipation of change in the frequency of therapeutic sessions, or the therapeutic focus over the duration of the trial.
   * Recent 2-month medication changes
5. Contraindication to receive TMS:

   * Cardiac pacemakers, implanted medication pumps, intracardiac lines, or acute, unstable cardiac disease.
   * Intracranial implant (e.g., aneurysm clips, shunts, stimulators, cochlear implants, stents, or electrodes) or any other metal object within or near the head, excluding the mouth, which cannot be safely removed.
   * Clinically significant abnormality or clinically significant unstable medical condition, as indicated by medical history, physical examination, ECG results, or clinical laboratory testing, that in the Investigator's judgment might pose a potential safety risk to the subject or limit interpretation of the trial results, e.g., any uncontrolled thyroid disorders, hepatic, cardiac, pulmonary and renal malfunctioning.
6. Women who are currently pregnant or not using a medically acceptable means of birth control and women who are breastfeeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2016-03; Primary Completion 2016-07 (Actual); Study Completion 2016-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard Weiner, MD, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- rTMS and Cognitive Behavior Therapy: Transcranial magnetic stimulation
  Cognitive behavioral therapy
Period: Overall Study
Arm/Group | rTMS and Cognitive Behavior Therapy
Started | 2
Completed | 0
Not Completed | 2
Not completed — Withdrawal by Subject | 2

BASELINE CHARACTERISTICS:
Arm/Group | rTMS and Cognitive Behavior Therapy
Number analyzed (Participants) | 2
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 2
  >=65 years | 0
Age, Continuous [Mean (Full Range); unit: years] | 51.5 [48 to 55]
Gender [Count of Participants; unit: Participants]
  Female | 1
  Male | 1
Region of Enrollment [Number; unit: participants]
  United States | 2

OUTCOME MEASURES:

1. Primary Outcome: Remission Rate, as Measured by Y-BOCS
Description: Remission is defined as end-point Yale-Brown Obsessive Compulsive Scale (Y-BOCS) score less than the value of 16.
Time Frame: 6 weeks
Measure: Number; unit: percentage of participants
Arm/Group | rTMS and Cognitive Behavior Therapy
Number analyzed (Participants) | 2
percentage of participants | 50

2. Secondary Outcome: Complete Response, as Measured by Y-BOCS
Description: Complete response is defined as a reduction of Y-BOCS score greater than 35%.
Time Frame: 6 weeks
Measure: Number; unit: percentage of participants
Arm/Group | rTMS and Cognitive Behavior Therapy
Number analyzed (Participants) | 2
percentage of participants | 50

3. Secondary Outcome: Partial Response Rate, as Measured by Y-BOCS
Description: Partial response is defined as a reduction of greater than 25%.
Time Frame: 6 weeks
Measure: Number; unit: percentage of participants
Arm/Group | rTMS and Cognitive Behavior Therapy
Number analyzed (Participants) | 2
percentage of participants | 50

4. Secondary Outcome: Percentage of Adverse Events
Time Frame: 6 weeks
Measure: Number; unit: percentage of adverse events
Arm/Group | rTMS and Cognitive Behavior Therapy
Number analyzed (Participants) | 2
percentage of adverse events | 0

ADVERSE EVENTS:
Arm/Group | rTMS and Cognitive Behavior Therapy
Serious Adverse Events (participants affected / at risk) | 0/2
Other Adverse Events (participants affected / at risk) | 0/2

LIMITATIONS AND CAVEATS:
This trial was terminated early leading to small numbers of subjects analyzed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes